CLINICAL TRIAL: NCT02546492
Title: Treatment of Chronic Antibody-mediated Rejection in Kidney Transplant With Acthar
Acronym: TGActhar
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow Enrollment
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Abdoleza Haririan, Medical director, Kidney and Pancreas Transplant Program, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00063872
Record Dates: First submitted 2015-04-10; First posted 2015-09-11 (Estimated); Results first posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Transplant Glomerulopathy
MeSH Terms: interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Acthar (Experimental): The study cohort. In this cohort Acthar gel will be administered to the enrolled patient with chrnic AMR.
  Interventions: Drug: Acthar gel

INTERVENTIONS:
Drug: Acthar gel — Administration of the study drug in addition to the current maintenance immunosuppressive agents
  Other Names: ACTH (Adrenocorticotropic hormone)

SUMMARY:
This is an open label safety and feasibility trial using Acthar® in addition to the investigators center-specific standard therapy, which could include increase in maintenance immunosuppression, high dose IVIG (intravenous immunoglobulin) (2 g/Kg), and/or Rituximab, in patients with chronic antibody-mediated rejection (CAMR).

DETAILED DESCRIPTION:
Subjects will receive Acthar® 40 units twice a week subcutaneously for 2 weeks. If the drug is well tolerated the dose will be increased to 80 units twice a week for another 22 weeks. The patients will be maintained on their center-specific standard maintenance regimen, typically consisting of Tacrolimus, mycephenolate mofetil/Sodium, and prednisone.

After screening for the inclusion/exclusion criteria, the patients will be consented and enrolled in the study. The initial visit and subsequent study-related visits at 4, 8, 12, 24, 36 and 52 weeks will include routine evaluation and physical examination and laboratory studies including CBC (complete blood count), electrolyte panel, eGFR, albumin, liver enzymes, and Calcineurin inhibitor (CNI)/sirolimus drug level, according to the center's standard of care. Donor-specific antibody (DSA) will be tested at week 24, and 52 and patients will undergo a biopsy at week 52, as a part of the investigators standard of care. The biopsies will be evaluated by light and electron microscopy using standard histological Banff criteria, and staining for CD68.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Morphologic diagnosis of CAMR, by light &/or electron microscopy any time after transplantation
* Current or previously documented donor-specific antibody (DSA) and/or focal or diffuse peritubular capillary C4d staining by immunohistochemistry
* eGFR>25 ml/min

Exclusion Criteria:

* Diagnosis of malignancy within a year prior to enrollment (except cured cutaneous basal cell or squamous cell carcinoma).
* Lack of evidence of antibody involvement
* Pregnancy, lactation, or refusal to use birth control in women of child bearing potential
* Active infection, or history of HIV
* History of liver or thoracic transplant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abdolreza Haririan, MD, MPH, Principal Investigator — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - University of Alabama School of Medicine, Alabama Transplant Center, Birmingham, Alabama
  - Unniversity of Maryland Medical Center, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Groups:
- Acthar: The study cohort. In this cohort Acthar gel will be administered to the enrolled patient with chronic antibody-mediated rejection (AMR).
  Acthar gel: Administration of the study drug in addition to the current maintenance immunosuppressive agents
Period: Overall Study
Arm/Group | Acthar
Started | 6
Completed | 1
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- All Participants Have Biopsy Proven Chronic Antibody Mediated Rejection, and Will Receive Acthar.: In this cohort Acthar gel will be administered to all the enrolled patient with chronic AMR.
  There is a single arm in this study.
  Acthar gel: Administration of the study drug in addition to the current maintenance immunosuppressive agents
Arm/Group | All Participants Have Biopsy Proven Chronic Antibody Mediated Rejection, and Will Receive Acthar.
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: Years] | 54.5 [33 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
eGFR (estimated Glomerular Filtration Rate) [Mean (Standard Deviation); unit: ml/min/1.73 m^2] | 49.2 (14.6)
Serum Creatinine [Mean (Standard Deviation); unit: mg/dl] | 1.75 (0.56)
Urine Albumin [Mean (Standard Deviation); unit: mg/L] | 745 (771.5)
Urine Albumin Creatinine Ratio [Mean (Standard Deviation); unit: mg/g Creatinine] | 722.8 (957.5)

OUTCOME MEASURES:

1. Primary Outcome: Safety (Serious Adverse Events)
Description: Participants will be monitored for Serious Adverse Events, as follows (as described in ClinicalTrials.gov) Death, Life-threatening events, Hospitalization (initial or prolonged), Disability and events that requires intervention to prevent permanent impairment or damage.
  Other (non serious) events which were anticipated or unanticipated (as described in ClinicaTrials.gov) will be monitored.
  ASSESSMENT: The subjects will be assessed at regular intervals through a questionnaire for Acthar related events, physician evaluation at clinical visits, and self reporting.
Time Frame: 12 months
Population: All participants were monitored for adverse events throughout their participation.
Measure: Count of Participants; unit: Participants
Groups:
- Serious Adverse Events (SAE): All study participants who received the study drug
Arm/Group | Serious Adverse Events (SAE)
Number analyzed (Participants) | 6
Participants | 2

2. Secondary Outcome: Efficacy Outcome
Description: composite of graft loss, death, decrease in eGFR>10%, and increase in proteinuria
Time Frame: 1 year
Population: Study participants who received the study drug
Measure: Count of Participants; unit: Participants
Groups:
- Efficacy Outcomes: 1 Death , 1 with decreased GFR>10%, 1 with increased proteinuria during the study period of one year
Arm/Group | Efficacy Outcomes
Number analyzed (Participants) | 6
Participants
  Composite outcome | 3
  Death | 1
  Decreased GFR>10% | 1
  Increased proteinuria | 1

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Participants Received Acthar: All participants in the study received Acthar.
Arm/Group | Participants Received Acthar
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Received Acthar (N=6)
Hospitalized (Renal and urinary disorders) | 1 (1)
Hospitalization (Endocrine disorders) | 1 (1) — New onset diabetes
Death (General disorders) | 1 (1) — Participant withdrew from the study due to general debility. He was found down (fallen)at home, medics pronounced him deceased, per report from spouse.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Received Acthar (N=6)
Cramps of hands and fingers (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness and Vertigo (Nervous system disorders) | 1 (1)
Tightness of Chest (Cardiac disorders) | 1 (1)
Weight gain (Metabolism and nutrition disorders) | 1 (1)
Irritablility (Nervous system disorders) | 1 (1)
Moon Face (Swelling of face) (Endocrine disorders) | 1 (1)
Elevated Blood Pressure (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Only one participant completed the treatment with the study drug Acthar (24 weeks). The other five (5) individuals withdrew from the study early, therefore we are not able to analyze/interpret the efficacy of the study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT02546492/Prot_SAP_000.pdf